# **Informed Consent Form (ICF)**

Effectiveness of
Individualized Dietary
Counseling and Nutritional
Monitoring in Reducing
Cancer-Associated Cachexia
among Female Breast Cancer
Patients
07 February 2024

#### **Informed Consent**

You are being invited to participate in a research study conducted at Fauji Foundation Hospital, Rawalpindi. The purpose of this study is to determine the effectiveness of individualized dietary counseling and nutritional monitoring in reducing cancer-associated cachexia among female patients with advanced breast cancer.

## **Purpose of the Study**

This study aims to evaluate if regular, personalized dietary counseling can reduce the severity of cachexia, a condition involving weight loss and muscle wasting, and improve your quality of life.

#### **Procedures**

If you choose to participate, you will be randomly assigned to one of two groups. One group will receive standard cancer care, and the other will receive additional nutritional counseling, dietary plans, and regular follow-ups every 15–21 days over six months.

#### **Potential Risks**

The risks associated with this study are minimal. You may experience minor discomfort during nutritional assessments, and there may be emotional responses to discussions about your health status.

#### **Potential Benefits**

You may benefit from personalized nutrition support, which could improve your physical health, nutritional status, and overall well-being. The findings may also benefit future patients.

## Confidentiality

All information collected will be kept strictly confidential. Your identity will not be revealed in any publication or presentation.

## **Voluntary Participation**

Your participation is voluntary. You can withdraw at any time without affecting your medical care or legal rights.

#### **Contact Information**

If you have any questions about this study, you may contact:

Dr Rida Maria

+92344-8804194

## **Consent Statement**

I have read and understood the information provided in this form. I have had the opportunity to ask questions, and all my questions have been answered to my satisfaction. I voluntarily agree to participate in this study.

| Participant's Name: | |
|---------------------------|-------|
| Participant's Signature: | Date: |
| Investigator's Name: | |
| Investigator's Signature: | Date: |